CLINICAL TRIAL: NCT00931996
Title: Clinical and Computational Studies of Dopamine Function in Schizophrenia
Brief Title: Oculomotor and Spatial Cognition Deficits in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to low accrual.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey R. Bishop, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2001-0522; R01MH062134 (NIH); R01MH080066 (NIH)
Record Dates: First submitted 2009-06-25; First posted 2009-07-02 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia; antipsychotic; risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Antipsychotic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antipsychotic (Experimental): Antipsychotic
  Interventions: Drug: Antipsychotic

INTERVENTIONS:
Drug: Antipsychotic — Risperidone is the first line antipsychotic followed by others per clinician choice. Flexible dosing QD x 4-6 weeks.

SUMMARY:
DESCRIPTION: (Verbatim from the Applicant's Abstract) Abnormalities of eye movement control and spatial cognition are well-established deficits in schizophrenia. However, the regional disturbances in brain function causing these deficits are not yet known. This application proposes a series of integrated behavioral studies designed to identify causes of deficits in schizophrenia.

DETAILED DESCRIPTION:
We will be assessing clinical symptoms and cognition before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Inclusion criteria for this study are (1) able and willing to give written informed consent; (2) no contraindications to MRI (cardiac pacemaker, aneurysm clip, cochlear implants, IUD, shrapnel, history of metal fragments in eyes, neurostimulators or other metal devices, weight of 250lbs or more, claustrophobia) and (3) medically stable. Sedation will not be used for MRI studies because cooperation is essential.

Exclusion Criteria:

* Any subject is excluded from the imaging studies if they have any contraindications to MRI such as cardiac pacemaker, aneurysm clip, cochlear implants, pregnancy in the later stages (because of body size and limited comfort for MRI studies), IUD, shrapnel, history of metal fragments in eyes, neurostimulators, weight of 250 lbs. or more, or claustrophobia. Individuals with mental retardation, neurologic disease or significant medical illness that might effect neuronal or vascular physiology will not be recruited.

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Sweeney, PhD, Principal Investigator — UIC/UTSW
Locations (1):
- UIC Center for Cognitive Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Antipsychotic: Antipsychotic treatment
Period: Overall Study
Arm/Group | Antipsychotic
Started | 12
Completed | 5
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Antipsychotic
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 11
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS) Score Change From Baseline.
Description: Positive and Negative Syndrome Scale (PANSS) Total Score. 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers. PANSS Total score minimum = 30, maximum = 210 Higher scores represent more severe symptoms. A positive change score (baseline-6 weeks) indicates an improvement in symptoms.
Time Frame: Baseline and 6 weeks
Population: Completers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antipsychotic
Number analyzed (Participants) | 5
units on a scale | 7.4 (12.9)

ADVERSE EVENTS:
Arm/Group | Antipsychotic
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antipsychotic (N=12)
EPS (Nervous system disorders) | 2 (2) — Extrapyramidal side effects assessed with Simpson Angus Rating Scale

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No